CLINICAL TRIAL: NCT04305574
Title: Getting it Right: Towards Responsible Social Media Use During a Pandemic
Brief Title: Social Media Use During COVID-19
Status: Completed | Type: Observational
Sponsor: Jean Liu (Other)
Responsible Party: Sponsor-Investigator, Jean Liu, Assistant Professor, Yale-NUS College
Organization: Yale-NUS College (Other)
Other Study IDs: 2020-CERC-001
Record Dates: First submitted 2020-03-08; First posted 2020-03-12 (Actual); Last update posted 2020-07-07 (Actual); Status verified 2020-07

CONDITIONS: Coronavirus; Depression; Anxiety; Stress
Keywords: COVID-19; Social media; Communication
MeSH Terms: conditions — Coronavirus Infections; Depression; Anxiety Disorders; COVID-19; Communication

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Community sample: We plan to recruit a representative sample of the Singapore population.
  Interventions: Behavioral: Use of social media during COVID-19

INTERVENTIONS:
Behavioral: Use of social media during COVID-19 — Participants' self-reported use of an official WhatsApp channel to receive and share news about COVID-19
  Other Names: WhatsApp

SUMMARY:
The investigators plan to conduct a cross-sectional survey to examine how social media use during COVID-19 relates to: (1) information management, (2) assessment of the situation, and (3) affect.

ELIGIBILITY:
Inclusion Criteria:

* At least 21 years
* Has stayed in Singapore for at least 2 years

Exclusion Criteria:

* Below 21 years
* Has stayed in Singapore for less than 2 years

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Representative sample of the Singapore population
Sampling Method: Non-Probability Sample
Enrollment: 1145 (Actual)
Dates: Start 2020-03-07 (Actual); Primary Completion 2020-04-21 (Actual); Study Completion 2020-04-21 (Actual)

PRIMARY OUTCOMES:
Depression, Anxiety and Stress Scale | Single measurement (upon study enrolment)
  21-item validated scale assessing symptoms of depression, anxiety, and stress (DASS-21): Min score = 0, Max score = 21; higher score indicates a worse outcome

OTHER OUTCOMES:
Assessment of COVID-19 situation | Single measurement (upon study enrolment)
  3 items on fear of the situation, confidence the government can manage the situation, and assessed chance of being infected (each rated using 4-point scales: min = 1, max = 4; higher scores indicate increased confidence / likelihood / fear)
Familiarity and trust in COVID-related rumours | Single measurement (upon study enrolment)
  Participants' self-report of their familiarity (yes/no) and belief of specific (yes/no), and whether they shared these on social media (yes/no)

CONTACTS AND LOCATIONS:
Overall Officials: Jean Liu, PhD, Principal Investigator — Yale-NUS College
Locations (1):
- Yale-NUS College, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No
Due to stipulations by the Institutional Review Board, data cannot be shared.

REFERENCES:
- [Derived] Liu JCJ, Tong EMW. The Relation Between Official WhatsApp-Distributed COVID-19 News Exposure and Psychological Symptoms: Cross-Sectional Survey Study. J Med Internet Res. 2020 Sep 25;22(9):e22142. doi: 10.2196/22142. PMID 32877349